CLINICAL TRIAL: NCT06569979
Title: The Knowledge Gaps of Amputee Rehabilitation Course Content in Physiotherapy Curriculum According to International Classification of Functioning, Disability and Health (ICF)
Brief Title: The Knowledge Gaps of Amputee Rehabilitation Course Content in Physiotherapy Curriculum
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Hatice Gül, Lecturer PhD, Akdeniz University
Other Study IDs: 202391-12/12/2023
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Amputation; Rehabilitation; ICF
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Academicians who continued to teach amputee rehabilitation in different higher education institutions in Turkey were included in the study.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The survey was developed using the Google Forms platform. The first part of the questionnaire consisted of descriptive information such as age, gender, duration of academic experience. In addition to this informations, the questionnaire also included information related the status of use ICF in any fields.
  In the other part of the questionnaire, a total of 59 questions (16 related to body functions, 3 related to body structures, 30 related to activity and participation, 10 related to environmental factors) were asked to the academicians whether these categories are present in the amputee rehabilitation course content. Academicians were asked to answer "yes" or "no" to each question.

SUMMARY:
Understanding the knowledge gaps of amputee rehabilitation course content is essential for addressing these gaps. Identifying the course contents according to International Classification of Functioning, Disability and Health (ICF) can be a starting point for determining the gaps. This study aimed to investigate which amputee-specific ICF categories are underemphasized in the course content.

DETAILED DESCRIPTION:
For understanding the knowledge gaps of amputee rehabilitation course content, a total of 59 amputee-specific ICF categories were asked to the academics whether these categories are present in the amputee rehabilitation course content. Academics were asked to answer "yes" or "no" to each question. Cochrane Q test was used to test for differences between the frequencies of ICF categories.

Sleep functions, high-level cognitive functions in the field of body functions, writing and handling stress in the activity sub-domain, most of the categories in the participation sub-domain and environmental factors were significantly underemphasized in the course content.This study identifies the knowledge gaps of amputee rehabilitation course content in physiotherapy curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Academicians who continued to teach amputee rehabilitation in different higher education institutions in Turkey were included in the study.

Exclusion Criteria:

* Individuals who did not teach the whole course but contributed to only a part of it were not included in the study

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Academicians aged 25-80 and continued to teach amputee rehabilitation in different higher education institutions in Turkey were included in the study.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Survey | 1 day
  The survey was developed using the Google Forms platform. The first part of the questionnaire consisted of descriptive information such as age, gender, duration of academic experience. In addition to this informations, the questionnaire also included information related the status of use ICF in any fields.
  In the other part of the questionnaire, a total of 59 questions (16 related to body functions, 3 related to body structures, 30 related to activity and participation, 10 related to environmental factors) were asked to the academicians whether these categories are present in the amputee rehabilitation course content. Academicians were asked to answer "yes" or "no" to each question.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Gül, Principal Investigator — Akdeniz University Vocational School of Health Services
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholten I, Barradell S, Bickford J, Moran M. Twelve tips for teaching the International Classification of Functioning, Disability and Health with a view to enhancing a biopsychosocial approach to care. Med Teach. 2021 Mar;43(3):293-299. doi: 10.1080/0142159X.2020.1789082. Epub 2020 Jul 9. PMID 32645280